CLINICAL TRIAL: NCT01648634
Title: A Randomized, Double-Blind, Placebo-Controlled, Multi-center Study to Examine the Effect of Nebivolol, a Beta-Blockade Drug, for the Prevention of Ventricular Systolic Dysfunction in Patients With Duchenne Muscular Dystrophy
Brief Title: Nebivolol for the Prevention of Left Ventricular Systolic Dysfunction in Patients With Duchenne Muscular Dystrophy
Acronym: NEBIDYS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Association Française contre les Myopathies (AFM), Paris (Other); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: P090202; 2010-020047-12 (EudraCT Number)
Record Dates: First submitted 2012-07-20; First posted 2012-07-24 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Duchenne Muscular Dystrophy; Cardiomyopathy; Heart Failure
Keywords: Nebivolol; beta-blockade treatment
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Cardiomyopathies; Heart Failure | interventions — Nebivolol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nebivolol (Experimental)
  Interventions: Drug: Nebivolol
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nebivolol — A 1.25mg-test dose will be administrated to assess the treatment tolerance before randomization. A forced titration of nebivolol will be performed with 2 weeks periods. Full dose of nebivolol is 5mg/day (7.5mg/day for patients whose weight is>60kg)
  Arms: Nebivolol
Drug: Placebo — A 1.25mg-test dose of nebivolol will be administrated to assess the treatment tolerance before randomization. A forced titration of placebo will be performed with 2 weeks periods. Full dose of placebo is 5mg/day (7.5mg/day for patients whose weight is>60kg)
  Arms: Placebo

SUMMARY:
The objective is to determine whether nebivolol, a beta-blockade drug, can prevent the development of heart disease in patients with Duchenne muscular dystrophy aged 10 to 15 year-old.

DETAILED DESCRIPTION:
A 1.25 mg-test dose will be administrated to assess the treatment tolerance before randomization. A forced titration of nebivolol and placebo will be performed with 2 weeks periods. Full dose of nebivolol and placebo is 5mg/day (7.5mg/day for patients whose weight is>60kg).

ELIGIBILITY:
Inclusion Criteria:

* Duchenne muscular dystrophy genetically proven
* Age between 10 and 15 years
* Left ventricular ejection fraction assessed by radionuclide angiography or echocardiography ≥50% and measured within 3 months
* Systolic blood pressure ≥80 mmHg
* Diastolic blood pressure ≥70 mmHg

Exclusion Criteria:

* Heart rate <50 bpm
* 2nd or 3rd degree atrioventricular blocks, sinus node dysfunction
* Asthma or bronchospasm
* Severe peripheral circulatory disease
* Hypersensitivity to nebivolol or excipients
* Metabolic acidosis
* Blood urea >7 mmol/l
* Liver transaminases enzymes >6 fold the upper limit of normal
* Formal indication for beta-blockade treatment
* Cardiac treatments except angiotensin-converting enzyme inhibitors
* Participation to another clinical trial within 3 months

Ages: 10 Years to 15 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2012-02-13 (Actual); Primary Completion 2021-07-20 (Actual); Study Completion 2021-07-20 (Actual)

PRIMARY OUTCOMES:
Left ventricular systolic dysfunction | at 5 years
  Development of left ventricular systolic dysfunction with an ejection fraction < 45%

SECONDARY OUTCOMES:
Right ventricular ejection fraction | at 5 years
  Right ventricular ejection fraction assessed by radionuclide angiography or echocardiography
NT-ProBNP | at 1, 2, 3, 4, and 5 years
  NT-ProBNP
Left ventricular dysfunction | at 10 years
  Development of left ventricular dysfunction
Hospitalizations | at 10 years
  hospitalizations for heart failure
Mortality | at 10 years ((5-years open label extension)
  Cardiovascular mortality

CONTACTS AND LOCATIONS:
Overall Officials: Henri-Marc BECANE, MD,PhD, Principal Investigator — Armand Trousseau Hospital
Locations (1):
- Armand Trousseau Hospital, Paris, France